CLINICAL TRIAL: NCT05251376
Title: A Phase 1, Single Dose, Open-label, Safety, Tolerability, and Pharmacokinetic Study of LYN-014 in Individuals With Opioid Use Disorder Who Are Stable on Methadone Therapy
Brief Title: Study of LYN-014 in Individuals With Opioid Use Disorder Who Are Stable on Methadone Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Lyndra Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYN-014-C-101; 4UH3DA050310-02 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Opioid Use Disorder, Moderate
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular | interventions — Methadone; Morphine; X-Rays; Radiography, Abdominal; Hematologic Tests; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LYN-014 Extended-Release Levomethadone HCl (Experimental): Extended-release levomethadone HCl 187 mg administered orally once on Day 8 of the study.
  Interventions: Drug: Levomethadone HCl; Drug: Methadone; Drug: Morphine Sulfate; Diagnostic Test: x-ray; Diagnostic Test: blood tests

INTERVENTIONS:
Drug: Levomethadone HCl — One dose given orally on Day 8 of the study.
  Other Names: extended-release levomethadone
Drug: Methadone — Daily usual oral dose given on Day 1 and Day 2 of the study.
  Other Names: oral methadone
Drug: Morphine Sulfate — Administered daily and as needed from Day 3 of the study until subject back on usual daily methadone dose.
  Other Names: morphine
Diagnostic Test: x-ray — Abdominal x-rays done at specific study timepoints to assess the location of the LYN-014.
  Other Names: abdominal x-ray
Diagnostic Test: blood tests — Done at specific timepoints throughout the study for PK (pharmacokinetics), genotyping and safety labs.
  Other Names: Blood draws, lab tests

SUMMARY:
A Phase 1, Single Dose, Open-label, Safety, Tolerability, and Pharmacokinetic Study of LYN-014 in Individuals with Opioid Use Disorder Who are Stable on Methadone Therapy

DETAILED DESCRIPTION:
Lyndra Therapeutics is currently developing extended release (ER) capsules for weekly administration across therapeutic areas with certain medications for which consistent pharmacokinetics (PK) or enhanced adherence may translate to improved efficacy, and possibly better safety. LYN-014 ER capsules are intended to provide comparable levomethadone exposure to daily treatment with racemic methadone for people with opioid use disorder (OUD). Compared to daily methadone dosing, LYN-014 could provide greater accessibility to methadone therapy and reduce the time devoted to obtaining medication the number of visits to methadone clinics, and thus reduce the stigma associated with methadone treatment, improve the quality of life for patients, and reduce the potential for diversion. This single dose study will evaluate the safety, tolerability, and PK of LYN-014 in individuals with OUD who are stable on daily methadone treatment. Data from this study will inform formulation optimization and dose selection for further development.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, individuals must meet all the following inclusion criteria at Screening (and at other timepoints, where specified):

Male or female aged ≥18 and ≤59 years. Body mass index of ≥18 kg/m2 and ≤33 kg/m2. Moderate or severe OUD according to the DSM-5 criteria. Clinically stable (for at least 6 months) on oral daily methadone therapy at a dose of 80 to 100 mg and have been taking the same dose for at least 3 months, and are stably engaged in a methadone program, confirmed by a methadone provider and defined as (1) demonstrates evidence of regular attendance, (2) has not had problems with missed visits, and (3) consistently demonstrates drug-negative urine samples (except for cannabis).

Agree to provide the study site with contact information for the clinic where they get methadone and agree that a study physician can contact the clinician providing methadone to confirm appropriateness for study participation and to manage their transition into the study and from the study back to their opioid treatment program.

Able to read and understand study procedures and provide written informed consent before the initiation of any protocol-specific procedures.

Willing to comply with all protocol-specified procedures and availability for the duration of the study (e.g., participant is not aware of any emergent life-changes or potential family emergencies that would interfere with a 40+ day inpatient stay).

Exclusion Criteria:

To be eligible to participate in the study, individuals must not meet any of the following exclusion criteria at Screening (and at other timepoints, where specified):

1. Known clinically significant esophageal or GI disease, including but not limited to:

a. Known strictures such as esophageal web, pyloric stenosis, small intestinal stricture, or individuals with high risk of stricture, ie, Crohn's disease b. Diagnosis of a condition known to elevate or lower gastric pH, eg, achlorhydria or hypochlorhydria c. Prior small or large bowel obstructions or varices d. Prior abdominal or upper GI surgery (prior uncomplicated laparoscopic procedures are permitted) e. History of dysphagia or aspiration in the last 5 years f. History of an esophageal motility disorder or undergoing treatment for a gastric motility disorder g. Significant history of diarrhea or constipation (non-methadone related) within 3 months of Screening h. Fewer than 3 bowel movements per week, on average i. Multiple episodes of abdominal pain in the prior 3 months j. Moderate or severe dysmenorrhea or menorrhagia (with use of pain medication) in the prior 3 months.

k. History of gastroparesis, rumination, autoimmune gastritis, H.pylori gastritis, or irritable bowel syndrome l. History compatible with acid reflux (heartburn, regurgitation, dysphagia, chest pain, water brash, globus sensation, odynophagia) m. Medical history compatible with Achlorhydria (i.e., history of autoimmune gastritis, pernicious anemia, H. plylori infection, partial gastrectomy).

1. History of moderate to severe Acid Reflux Disease or a score of ≥2 on the Acid Reflux Severity Scale (ARSS), indicating moderate to severe symptoms. The ARSS scale is as follows:

   None = 0 no symptoms Mild = 1 awareness of symptom, but easily tolerated Moderate = 2 discomfort sufficient to cause interference with normal activities Severe = 3 incapacitating, with inability to perform normal activities.
2. Individuals with PILL 5 swallowing questionnaire score of 5 or greater.
3. Medical history or current diagnoses indicating the presence of any of the following conditions:

   1. Presence of an uncontrolled, unstable, or clinically significant medical condition, mental impairment, or psychiatric disease (e.g., schizophrenia, bipolar, major depression, or borderline personality disorder) that could put the subject at risk because of participation in the study, interfere with the subject's ability to participate in the study or influence the interpretation of safety or PK evaluations
   2. History of a major cardiovascular event (myocardial infarction, cardiac surgery or revascularization, unstable angina, stroke, or transient ischemic attack) or a hospitalization for heart failure within 6 months of Screening
   3. Presence of Long QT Syndrome
   4. Any clinically significant illness, medical or surgical procedure or trauma within 4 weeks of Screening, in the opinion of the Sponsor/designee or Principal Investigator
   5. Known immunocompromised status, including individuals who have undergone organ transplantation, on immunosuppression for an immune mediated disease, or are positive for HIV
   6. Positive test for active hepatitis B at Screening, unless hepatitis B infection has been resolved for ≥1 year
   7. Donated more than 250 mL of blood within 4 weeks of Screening
   8. Difficulties with venipuncture/cannulation, including difficulty accessing veins for blood sampling and/or history of coagulopathy or endocarditis
   9. Suicidal ideation associated with actual intent and a method or plan in the past 6 months, as measured by the C-SSRS (i.e., "Yes" answers on items 4 or 5) at Screening or Day 1, or has a history of suicide attempt within the last 2 years
   10. Chronic pain that requires chronic opioid treatment
   11. Active SARS-CoV-2 infection, as defined in the site-specific COVID 19 Risk Mitigation Plan
   12. History of pernicious anemia
   13. History of advanced cirrhosis
4. Use of the below in the 2 weeks before enrollment:

   1. Proton pump inhibitors and H2 blockers
   2. Prokinetics
   3. Grapefruit juice, blood oranges, Seville (bitter) oranges, and star fruit
   4. Medications that may interfere with the absorption, metabolism, or excretion of methadone (see Appendix 18.1)
   5. Medications that have a known risk of Torsades des Pointes (see Appendix 18.2)
   6. Concomitant medications, natural remedies, supplements, or vitamins that are associated with changes to gastric motility or pH. Use of antacids is permissible, except for within 2 hours of dosing with LYN 014
   7. Benzodiazepines except for treatment of insomnia (short/medium acting benzodiazepines used occasionally (1 or 2 times per week)
   8. Hormonal contraceptives
5. Use of blood products within 3 months of Screening.
6. Medical history or current diagnosis of chronic obstructive pulmonary disorder, restrictive lung disease, asthma, or any condition that could contribute to respiratory distress during study participation.
7. Clinically significant abnormal safety (e.g., physical examination, vital signs) or safety laboratory assessments at Screening, specifically:

   1. Presence of a clinically significant abnormal laboratory result on blood or urine safety tests
   2. Anemia (hemoglobin below lower limit of normal reference range and considered to be clinically significant)
   3. Alanine aminotransferase or aspartate aminotransferase ≥3.0 × upper limit of normal or total bilirubin ≥1.5 × upper limit of normal
   4. Moderate or severe renal insufficiency (Glomerular Filtration Rate <60 mL/min as determined using the Cockcroft Gault formula)
   5. Heart rate <60 beats per minute (bpm)
   6. Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
   7. Glycated hemoglobin (hemoglobin A1c; HbA1c) ≥6.5 mmol/L
   8. Thrombocytopenia (platelets <150 × 109/L) or bleeding diathesis (International Normalization Ratio > 1.4)
   9. Positive fecal occult blood test (FOBT) at Screening
8. The following specified patterns of substance use:

   1. Concomitant substance use disorder other than OUD, caffeine use disorder, or nicotine use disorder
   2. Positive urine drug screen for cocaine, amphetamine, methamphetamine, barbiturates, propoxyphene, phencyclidine, or buprenorphine
   3. Cannabis use disorder
   4. Positive ethanol breathalyzer result
9. Women of childbearing potential and men, who are unwilling to use acceptable means of contraception through the EOS. For clarity, women who are at least 1 year post menopausal are considered not of childbearing potential and can be included in the study. Acceptable means of contraception include:

   1. Individuals who have been surgically sterilized
   2. Females of childbearing potential: diaphragm, contraceptive sponge, or intrauterine device in use before enrollment, in combination with use of a condom for their male partners
   3. Males: condom in combination with any of the above means of contraception for their female partners
   4. All individuals: abstinence is only acceptable if a subject chooses not to be sexually active
10. Individuals who are nursing or have a positive or indeterminate pregnancy test at Screening (serum test) or Day 1 (urine test).
11. Use of any experimental agent within 3 months or 5 half lives of Screening, whichever is longer.
12. Employees or immediate family members of employees of the site, Sponsor, or study related vendors.
13. History of a serious allergic or hypersensitivity reaction to LYN 014 components or any components of morphine sulfate or ancillary medications.
14. History of X ray, computed tomography scan or angiogram of the abdomen within 1 year of Screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the LYN-014 dose when administered orally as a single dose | 52 days
  Incidence of treatment-emergent adverse events and serious adverse events
To characterize the PK of levomethadone for LYN-014 (Cmin) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate Cmin (minimum concentration)
To characterize the PK of levomethadone for LYN-014 (Tmin) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate Tmin (Time at minimum concentration)
To characterize the PK of levomethadone for LYN-014 (Cmax) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate Cmax (maximum concentration)
To characterize the PK of levomethadone for LYN-014 (Tmax) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate Tmax (Time at maximum concentration)
To characterize the PK of levomethadone for LYN-014 (Kel) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate Kel (Elimination Rate Constant)
To characterize the PK of levomethadone for LYN-014 (AUC0-20) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-20 (Area under the curve from 0-24 hours)
To characterize the PK of levomethadone for LYN-014 (AUC0-t) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-t (Area under the curve from 0 to t hours)
To characterize the PK of levomethadone for LYN-014 (AUC0-∞t) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-∞t (Area under the curve from 0 to infinity)
To characterize the PK of levomethadone for LYN-014 (C last) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate C last (Last measurable concentration)
To characterize the PK of levomethadone for LYN-014 (T last) | 52 days
  PK of levomethadone after oral administration of LYN-014, to include where possible and appropriate T last (Time at last measurable concentration)

SECONDARY OUTCOMES:
To characterize the PK of methadone enantiomers after methadone dosing (Cmin) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Cmin (Minimum Concentration)
To characterize the PK of methadone enantiomers after methadone dosing (Tmin) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Tmin (Time at minimum concentration)
To characterize the PK of methadone enantiomers after methadone dosing (Cmax) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Cmax (Maximum concentration)
To characterize the PK of methadone enantiomers after methadone dosing (Tmax) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Tmax (Time at maximum concentration)
To characterize the PK of methadone enantiomers after methadone dosing (Kel) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Kel (Elimination Rate Constant)
To characterize the PK of methadone enantiomers after methadone dosing (AUC0-24) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate AUC0-24 (Area under the curve from 0 to 24 hours)
To characterize the PK of methadone enantiomers after methadone dosing (AUC0-t) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate AUC0-t (Area under the curve from 0 to t hours)
To characterize the PK of methadone enantiomers after methadone dosing (AUC0-∞) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate AUC0-∞ (Area under the curve from 0 to infinity)
To characterize the PK of methadone enantiomers after methadone dosing (Clast) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Clast (Last measurable concentration)
To characterize the PK of methadone enantiomers after methadone dosing (Tlast) | 52 days
  PK of levomethadone and dextromethadone (S-enantiomer of methadone) after oral administration of methadone, to include where possible and appropriate Tlast (Time at last measurable concentration)
To characterize the PK of LYN 014 compared with that of daily methadone Cmax Extended Release to Cmax Immediate Release | 52 days
  Compare the PK ratio of Cmax (maximum concentration) ER (LYN-014) to Cmax (maximum concentration) IR (methadone).
To evaluate possible conversion of Levomethadone to Dextromethadone (Cmin) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Cmin (minimum concentration)
To evaluate possible conversion of Levomethadone to Dextromethadone (Tmin) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Tmin (Time at minimum concentration)
To evaluate possible conversion of Levomethadone to Dextromethadone (Cmax) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Cmax (Maximum concentration)
To evaluate possible conversion of Levomethadone to Dextromethadone (Tmax) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Tmax (Time at maximum concentration)
To evaluate possible conversion of Levomethadone to Dextromethadone (Kel) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Kel (elimination rate constant)
To evaluate possible conversion of Levomethadone to Dextromethadone (AUC0-24) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-24 (Area under the curve from 0 to 24 hours)
To evaluate possible conversion of Levomethadone to Dextromethadone (AUC0-t) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-t (Area under the curve from 0 to t hours)
To evaluate possible conversion of Levomethadone to Dextromethadone (AUC0-∞) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate AUC0-∞ (Area under the curve from 0 to infinity)
To evaluate possible conversion of Levomethadone to Dextromethadone (Clast) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Clast (last measurable concentration)
To evaluate possible conversion of Levomethadone to Dextromethadone (Tlast) | 52 days
  PK of dextromethadone after oral administration of LYN-014, to include where possible and appropriate Tlast (Time at last measurable concentration)
To assess gastrointestinal (GI) transit and exit properties of LYN 014. | 52 days
  GI transit and exit properties of LYN 014 assessed by X ray imaging and fecal recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Scranton, MD, MPH, Principal Investigator — Lyndra Therapeutics INC

IPD SHARING:
Plan to Share IPD: No